CLINICAL TRIAL: NCT02872012
Title: Cryoanesthesia for Intravitreal Injections
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Anjali Shah, Instructor in Ophthalmology and Visual Sciences, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00105826
Record Dates: First submitted 2016-06-02; First posted 2016-08-18 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Ocular Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Device: Yes

ARMS (6):
- Cryoanesthesia Device -5 degrees Celsius for 10 seconds (Experimental): All patients will have one eye randomized to receiving anesthesia via the cryoanesthesia device which anesthetizes by chilling rather than by use of drug, prior to receiving an intravitreal injection.
  Comment: Cryoanesthesia Device is the name of the device.
  Interventions: Device: Cryoanesthesia device
- Cryoanesthesia Device -5 degrees Celsius for 20 seconds (Experimental): All patients will have one eye randomized to receiving anesthesia via the cryoanesthesia device which anesthetizes by chilling rather than by use of drug, prior to receiving an intravitreal injection.
  Comment: Cryoanesthesia Device is the name of the device.
  Interventions: Device: Cryoanesthesia device
- Cryoanesthesia Device -7 degrees Celsius for 20 seconds (Experimental): All patients will have one eye randomized to receiving anesthesia via the cryoanesthesia device which anesthetizes by chilling rather than by use of drug, prior to receiving an intravitreal injection.
  Comment: Cryoanesthesia Device is the name of the device.
  Interventions: Device: Cryoanesthesia device
- Cryoanesthesia Device -10 degrees Celsius for 10 seconds (Experimental): All patients will have one eye randomized to receiving anesthesia via the cryoanesthesia device which anesthetizes by chilling rather than by use of drug, prior to receiving an intravitreal injection.
  Comment: Cryoanesthesia Device is the name of the device.
  Interventions: Device: Cryoanesthesia device
- Cryoanesthesia Device -10 degrees Celsius for 20 seconds (Experimental): All patients will have one eye randomized to receiving anesthesia via the cryoanesthesia device which anesthetizes by chilling rather than by use of drug, prior to receiving an intravitreal injection.
  Comment: Cryoanesthesia Device is the name of the device.
  Interventions: Device: Cryoanesthesia device
- Lidocaine (Active Comparator): Participants randomized to this arm will have their other eye receive anesthesia via the current standard of care treatment method (lidocaine) prior to receiving an intravitreal injection.
  Lidocaine: Lidocaine will be applied to the non-cryoanesthesia eye.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Device: Cryoanesthesia device — The study will be carried out in patients receiving bilateral injections. One eye will be anesthetized using the cryoanesthesia device, developed at the University of Michigan. This has been assessed to be a Non-significant Risk device.
  Arms: Cryoanesthesia Device -10 degrees Celsius for 10 seconds; Cryoanesthesia Device -10 degrees Celsius for 20 seconds; Cryoanesthesia Device -5 degrees Celsius for 10 seconds; Cryoanesthesia Device -5 degrees Celsius for 20 seconds; Cryoanesthesia Device -7 degrees Celsius for 20 seconds
Drug: Lidocaine — Lidocaine applied to the non-cryoanesthesia eye.
  Arms: Lidocaine

SUMMARY:
The cryoanesthesia (CA) device is designed to provide anesthesia to a focal area on the surface of the eye immediately prior to intraocular injections.

The investigators plan to carry out a pilot study to collect preliminary data on the effectiveness of the cryoanesthesia (CA) device in minimizing the pain caused by intravitreal injections (IVT).

ELIGIBILITY:
Inclusion Criteria:

* Bilateral macular disease due to either exudative macular degeneration or diabetic retinopathy requiring bilateral intravitreal injections
* Have had at least one prior intravitreal injection
* Able to give informed consent

Exclusion Criteria:

* Unilateral disease
* Unable to provide consent
* Preexisting conjunctival, episcleral or scleral defects or disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali R Shah, MD, Principal Investigator — Instructor in Ophthalmology and Visual Sciences
Locations (1):
- Kellogg Eye Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Besirli CG, Smith SJ, Zacks DN, Gardner TW, Pipe KP, Musch DC, Shah AR. Randomized Safety and Feasibility Trial of Ultra-Rapid Cooling Anesthesia for Intravitreal Injections. Ophthalmol Retina. 2020 Oct;4(10):979-986. doi: 10.1016/j.oret.2020.04.001. Epub 2020 Apr 15. PMID 32446842

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 participants were recruited. Each participant received 1 cryoanesthesia intervention in one eye and one standard of care lidocaine intervention in their other eye.
Groups:
- Cryoanesthesia Device -5 Degrees Celsius for 10 Seconds; Cryoanesthesia Device -5 Degrees Celsius for 20 Seconds; Cryoanesthesia Device -7 Degrees Celsius for 20 Seconds; Cyroanesthesia Device -10 Degrees Celsius for 10 Seconds; Cryoanesthesia Device -10 Degrees Celsius for 20 Seconds: All patients will have one eye randomized to receiving anesthesia via the cryoanesthesia device which anesthetizes by chilling rather than by use of drug, prior to receiving an intravitreal injection. Their other eye will receive anesthesia via the active comparator, lidocaine.
  Comment: Cryoanesthesia Device is the name of the device.
  Cryoanesthesia device: The study will be carried out in patients receiving bilateral injections. One eye will be anesthetized using the cryoanesthesia device, developed at the University of Michigan. This has been assessed to be a Non-significant Risk device.
  Patients will receive the cryoanesthesia at a temperature of -5C for 10 seconds, -5C for 20 seconds, 0C for 20 seconds, or -10C for 10 seconds.
Period: Overall Study
Arm/Group | Cryoanesthesia Device -5 Degrees Celsius for 10 Seconds | Cryoanesthesia Device -5 Degrees Celsius for 20 Seconds | Cryoanesthesia Device -7 Degrees Celsius for 20 Seconds | Cyroanesthesia Device -10 Degrees Celsius for 10 Seconds | Cryoanesthesia Device -10 Degrees Celsius for 20 Seconds
Started | 4 | 7 | 4 | 3 | 5
Completed | 3 | 7 | 4 | 3 | 5
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cryoanesthesia Device -10 Degrees Celsius for 10 Seconds; Cryoanesthesia Device -10 Degrees Celsius for 20 Seconds: All patients will have one eye randomized to receiving anesthesia via the cryoanesthesia device which anesthetizes by chilling rather than by use of drug, prior to receiving an intravitreal injection. Their other eye will receive anesthesia via the active comparator, lidocaine.
  Comment: Cryoanesthesia Device is the name of the device.
  Cryoanesthesia device: The study will be carried out in patients receiving bilateral injections. One eye will be anesthetized using the cryoanesthesia device, developed at the University of Michigan. This has been assessed to be a Non-significant Risk device.
  Patients will receive the cryoanesthesia at a temperature of -5C for 10 seconds, -5C for 20 seconds, 0C for 20 seconds, or -10C for 10 seconds.
- Total: Total of all reporting groups
Arm/Group | Cryoanesthesia Device -5 Degrees Celsius for 10 Seconds | Cryoanesthesia Device -5 Degrees Celsius for 20 Seconds | Cryoanesthesia Device -7 Degrees Celsius for 20 Seconds | Cryoanesthesia Device -10 Degrees Celsius for 10 Seconds | Cryoanesthesia Device -10 Degrees Celsius for 20 Seconds | Total
Number analyzed (Participants) | 3 | 7 | 4 | 3 | 5 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 2 | 1 | 3 | 9
  >=65 years | 1 | 6 | 2 | 2 | 2 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 3 | 2 | 2 | 16
  Male | 1 | 0 | 1 | 1 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Injection Pain
Description: Immediately after receiving the intravitreal injection, patient's will be asked to rate their pain on the Visual Analogue (Pain) Scale. The scale ranges from 0 to 10. 0 meaning no pain and 10 meaning the worst possible pain.
Time Frame: Immediately following the intravitreal injection
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Cyroanesthesia Device -5 Degrees Celsius for 20 Seconds; Cryoanesthesia Device -7 Degrees Celsius for 20 Seconds; Cryoanesthesia Device -10 Degrees Celsius for 10 Seconds; Cryoanesthesia Device -10 Degrees Celsius for 20 Seconds: All patients will have one eye randomized to receiving anesthesia via the cryoanesthesia device which anesthetizes by chilling rather than by use of drug, prior to receiving an intravitreal injection. Their other eye will receive anesthesia via the active comparator, lidocaine.
  Comment: Cryoanesthesia Device is the name of the device.
  Cryoanesthesia device: The study will be carried out in patients receiving bilateral injections. One eye will be anesthetized using the cryoanesthesia device, developed at the University of Michigan. This has been assessed to be a Non-significant Risk device.
  Patients will receive the cryoanesthesia at a temperature of -5C for 10 seconds, -5C for 20 seconds, 0C for 20 seconds, or -10C for 10 seconds.
- Standard of Care: Lidocaine: Participants randomized to this arm will have their other eye receive anesthesia via the current standard of care treatment method (lidocaine) prior to receiving an intravitreal injection.
  Lidocaine: Lidocaine will be applied to the non-cryoanesthesia eye.
Arm/Group | Cryoanesthesia Device -5 Degrees Celsius for 10 Seconds | Cyroanesthesia Device -5 Degrees Celsius for 20 Seconds | Cryoanesthesia Device -7 Degrees Celsius for 20 Seconds | Cryoanesthesia Device -10 Degrees Celsius for 10 Seconds | Cryoanesthesia Device -10 Degrees Celsius for 20 Seconds | Standard of Care: Lidocaine
Number analyzed (Participants) | 3 | 7 | 4 | 3 | 5 | 22
units on a scale | 7.0 (1.5) | 3.1 (0.6) | 3.0 (1.1) | 1.8 (0.8) | 2.4 (0.8) | 2.3 (0.4)

ADVERSE EVENTS:
Time Frame: 7 days after treatment
Groups:
- Cryoanesthesia Device -5 Degrees Celsius for 20 Seconds; Cryoanesthesia Device -7 Degrees Celsius for 20 Seconds; Cryoanesthesia Device -10 Degrees Celsius for 10 Seconds; Cryoanesthesia Device -10 Degrees Celsius for 20 Seconds: All patients will have one eye randomized to receiving anesthesia via the cryoanesthesia device which anesthetizes by chilling rather than by use of drug, prior to receiving an intravitreal injection.
  Comment: Cryoanesthesia Device is the name of the device.
  Cryoanesthesia device: The study will be carried out in patients receiving bilateral injections. One eye will be anesthetized using the cryoanesthesia device, developed at the University of Michigan. This has been assessed to be a Non-significant Risk device.
  Patients will receive the cryoanesthesia at a temperature of -5C for 10 seconds, -5C for 20 seconds, -7C for 20 seconds, -10C for 10 seconds, or -10C for 20 seconds.
- Standard of Care: Lidocaine Gel: Participants randomized to this arm will have their other eye receive anesthesia via one current standard of care treatment method (lidocaine gel) prior to receiving an intravitreal injection.
  Lidocaine gel: Lidocaine gel applied to the non-cryoanesthesia eye.
Arm/Group | Cryoanesthesia Device -5 Degrees Celsius for 10 Seconds | Cryoanesthesia Device -5 Degrees Celsius for 20 Seconds | Cryoanesthesia Device -7 Degrees Celsius for 20 Seconds | Cryoanesthesia Device -10 Degrees Celsius for 10 Seconds | Cryoanesthesia Device -10 Degrees Celsius for 20 Seconds | Standard of Care: Lidocaine Gel
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 0/4 | 0/3 | 0/5 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/7 | 0/4 | 0/3 | 0/5 | 0/22
Other Adverse Events (participants affected / at risk) | 0/3 | 0/7 | 0/4 | 0/3 | 0/5 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT02872012/Prot_000.pdf